CLINICAL TRIAL: NCT02406339
Title: Analysis of the Effectiveness of Neuromuscular Electrical Stimulation Associated to Vascular Occlusion in Functional Performance and Muscle Hypertrophy in Athlete's Basketball of High Performance. Blind Randomized Clinical Trial
Brief Title: Effectiveness of NMES Associated to Vascular Occlusion in Functional Performance and Muscle Hypertrophy in Athlete's
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Sao Paulo (Other)
Responsible Party: Principal Investigator, Rinaldo Roberto de Jesus Guirro, PhD, University of Sao Paulo
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: U1111-1143
Record Dates: First submitted 2015-03-14; First posted 2015-04-02 (Estimated); Last update posted 2017-07-21 (Actual); Status verified 2017-07

CONDITIONS: Electric Stimulation Therapy; Muscle Strength
Keywords: Physical Therapy; Rehabilitation; Neuromuscular Electrical Stimulation; Muscle Strength

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Control (No Intervention): Are not subject to any intervention.
- Electrotherapy (Experimental): The athletes will be submitted to NMES of bilateral quadriceps. The stimulation will be held in order to induce the move flexion / extension involuntary knee in extension machine, with resistance of 30% of maximum voluntary strength.
  Interventions: Device: NMES
- Electrotherapy + Vascular Occlusion (Experimental): The same as in Electrotherapy group, athletes are subjected to NMES associated total vascular occlusion of the members below the level of the groin.
  Interventions: Device: NMES; Device: Vascular Occlusion

INTERVENTIONS:
Device: NMES — Neuromuscular Electrical Stimulation
  Arms: Electrotherapy; Electrotherapy + Vascular Occlusion
Device: Vascular Occlusion — Restriction of sanguine flow to the lower limbs
  Arms: Electrotherapy + Vascular Occlusion

SUMMARY:
This study evaluates the effect of training with neuromuscular electrical stimulation (NMES) associated with vascular occlusion of the lower limbs, for increased strength and hypertrophy of the quadriceps muscle of professional basketball athletes.

DETAILED DESCRIPTION:
The pre-season preparation is seen as vital to maximize sports performance. However, there has been much debate on what the best strategy to prepare for use. Basketball is a sports activity of high intensity and volume of jumps, which are generally likely to cause injuries resulting from muscle imbalance and dynamic overload. Primarily in activities with eccentric contraction of the knee extensor muscles. A means of preventing injuries and optimization of sports performance is through strength training. Neuromuscular electrical stimulation (NMES) has been a physical therapy effective in increasing the recruitment of muscle fibers and strength. Another method that has been shown effective in increasing strength and muscle hypertrophy is the association of low intensity training and peripheral vascular occlusion. Therefore, the purpose of this study is to evaluate the effectiveness of neuromuscular electrical stimulation associated to vascular occlusion of lower limb muscle recruitment, strength and muscle hypertrophy. This will be met recruited basketball athletes of high performance, the males, aged between 18 and 30 years and BMI between 20 and 24 Kg/m2. The athletes will be randomized into four groups: group control (n = 15), group electrotherapy (n = 15) and group electrotherapy + vascular occlusion (n = 15). Will be carried out 12 sessions of treatment during the pre-season, and the volunteers evaluated before and after the pre-season and in middle the season, through the following instruments: Isokinetic Dynamometer, Surface Electromyography, Force Platform, Cross Section Area of Muscle, Vertical Jump, Functional Evaluation (Jump, Agility and Balance), Infrared Thermography and Numeric Scale of Pain Evaluation. For data analysis, normality test is used to verify the data distribution and consistent statistical test for the appropriate comparisons within and between groups, and thus considered two factors in the comparisons, time and group. Will adopt a significance level of 5%.

ELIGIBILITY:
Inclusion Criteria:

* The categories Basketball Athletes sub- 19, 21 and professional
* BMI between 20 and 24 kg / m²;
* To present physical and cardiorespiratory fitness, attested by the medical responsible for the team, for conducting evaluations and physical training;

Exclusion Criteria:

* Previous disease of circulatory order, nervous, metabolic, rheumatic and orthopedic; history of pain or muscle or joint injuries in the lower limbs in the last three months; subjects suffering from muscle fatigue complaint at the time of testing; athletes require the use of stabilizers to perform the tests;
* To present ankle instability assessed by questionnaire Foot and Ankle Outcome Score

Ages: 16 Years to 36 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 45 (Actual)
Dates: Start 2014-07 (Actual); Primary Completion 2017-03 (Actual); Study Completion 2017-05 (Actual)

PRIMARY OUTCOMES:
Analysis of muscle strength through isokinetic dynamometer (N / M). | 12 weeks
  The association of NMES and vascular occlusion of the lower limbs increases the isokinetic torque?
Analysis of hypertrophy through the cross section area of the muscle via ultrasound (mm). | 12 weeks
  The association of NMES and vascular occlusion of the lower limbs increases the cross-sectional area of the muscle?

SECONDARY OUTCOMES:
Analysis of GH Level by blood test (mg / L) | 12 weeks
  The association of NMES and vascular occlusion of the lower limbs increases the growth hormone (GH) levels after training?
Analysis of IGF-1 Level by blood test (mg / L) | 12 weeks
  The association of NMES and vascular occlusion of the lower limbs increases the insulin like growth factor-1 (IGF-1) after training?
Analysis of Star Excursion Balance Test (cm) | 12 weeks
  The association of NMES and vascular occlusion of the lower limbs improves balance of the athletes?
Performance Analysis in Illinois agility test (Time in seconds) | 12 weeks
  The association of NMES and vascular occlusion of the lower limbs improves agility of the athletes?
Muscle electromyographic analysis through the median frequency (Hz) and root mean square (RMS) | 12 weeks
  The association of NMES and vascular occlusion of the lower limbs increases the muscle activation and recruitment?

CONTACTS AND LOCATIONS:
Locations (1):
- Rinaldo Roberto de Jesus Guirro, Ribeirão Preto, São Paulo, Brazil